CLINICAL TRIAL: NCT02911844
Title: Estrogen Receptor Antagonist in Patients With Pulmonary Arterial Hypertension
Acronym: ERA-PAH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 824861
Record Dates: First submitted 2016-09-19; First posted 2016-09-22 (Estimated); Results first posted 2019-12-09 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-12

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Fulvestrant (Other): 500 mg administered intramuscularly (as two 5 mL injections) on days 0, 14, 28 and 56
  Interventions: Drug: Fulvestrant

INTERVENTIONS:
Drug: Fulvestrant — Fulvestrant 500 mg administered intramuscularly into the buttocks slowly as two 5 mL injections, one in each buttock, on days 0, 14, 28 and 56. Fulvestrant 250 mg (one 5 mL injection) will be used in patients with Child-Pugh Class B liver disease.
  Other Names: Faslodex

SUMMARY:
The main purpose of this clinical trial is to examine the feasibility and effects of fulvestrant in post-menopausal women with pulmonary arterial hypertension (PAH). The study will evaluate how well the drug is tolerated. The study will evaluate changes in circulating hematopoietic progenitor cells, plasma hormone levels, NT-proBNP, and other plasma biomarkers after the administration of fulvestrant. Changes in tricuspid annular plane systolic excursion, stroke volume index, right ventricular fractional area change, and other echo parameters after fulvestrant administration will be evaluated as well as changes in distance walked in six minutes.

ELIGIBILITY:
Inclusion Criteria:

* Previous documentation of mean pulmonary artery pressure > 25 mm Hg with a pulmonary capillary wedge pressure (or left ventricular end-diastolic pressure) < 16 mm Hg and pulmonary vascular resistance > 3 WU at any time before study entry.
* Diagnosis of PAH which is idiopathic, heritable, drug- or toxin-induced, or associated with connective tissue disease, congenital heart disease, portal hypertension, or HIV infection.
* Most recent pulmonary function tests with FEV1/FVC >50% AND either a) total lung capacity > 70% predicted or b) total lung capacity between 60% and 70% predicted with no more than mild interstitial lung disease on computerized tomography scan of the chest.
* Female, post-menopausal state, defined as:
* > 50 years old and a) have not menstruated during the preceding 12 months or b) have follicle-stimulating hormone (FSH) levels > 40 IU/L or
* < 50 years and FSH > 40 IU/L or
* having had a bilateral oophorectomy.
* Informed consent.

Exclusion Criteria:

* Age < 18.
* Treatment with estrogen or anti-hormone therapy (tamoxifen, anastrozole, etc.)
* WHO Class IV functional status.
* History of breast cancer.
* Clinically significant untreated sleep apnea.
* Left-sided valvular disease (more than moderate mitral valve stenosis or insufficiency or aortic stenosis or insufficiency), pulmonary artery or valve stenosis, or ejection fraction < 45% on echocardiography.
* Initiation of PAH therapy (prostacyclin analogues or receptor agonists, endothelin-1 receptor antagonists, phosphodiesterase-5 inhibitors, soluble guanylate cyclase stimulators) within three months of enrollment; the dose must be stable for at least 3 months prior to Baseline Visit. PAH therapy which is stopped and then restarted or has dose changes which are not related to initiation and uptitration will be allowed within 3 months prior to the Baseline Visit.
* Hormone therapy.
* Use of warfarin or other anticoagulant (use of aspirin is permitted).
* Platelet count <100,000.
* Renal failure (creatinine >/= 2.0).
* Child-Pugh Class C cirrhosis.
* Current or recent (< 6 months) chronic heavy alcohol consumption.
* Current use of another investigational drug (non-FDA approved) for PAH.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-04-10 (Actual); Primary Completion 2018-12-05 (Actual); Study Completion 2018-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven M Kawut, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Kawut SM, Pinder D, Al-Naamani N, McCormick A, Palevsky HI, Fritz J, Smith KA, Mazurek JA, Doyle MF, MacLean MR, DeMichele A, Mankoff DA. Fulvestrant for the Treatment of Pulmonary Arterial Hypertension. Ann Am Thorac Soc. 2019 Nov;16(11):1456-1459. doi: 10.1513/AnnalsATS.201904-328RL. No abstract available. PMID 31314997

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fulvestrant
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Fulvestrant
Number analyzed (Participants) | 5
Age, Continuous [Median (Full Range); unit: years] | 55 [52 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5
Childs-Pugh Class [Count of Participants; unit: Participants] — Child-Pugh Class consists of five clinical features and is used to assess the prognosis of chronic liver disease and cirrhosis. There are three distinct classes of increasing severity (A, B and C). Class is determined based on a score that accounts for five factors: total bilirubin level, serum albumin, INR, degree of ascites, and degree of hepatic encephalopathy. Class A is considered the best and indicates mild liver disease, Class B is moderate liver disease, and Class C is severe liver disease.
  Participants
    A | 5
    B or C | 0
World Health Organization functional class [Count of Participants; unit: Participants] — Classification based on evaluation of the participant.
  Class I: Patients without limitation of physical activity. Ordinary physical activity does not cause undue dyspnea or fatigue, chest pain or near-syncope.
  Class II: Patients with slight limitation of physical activity. They are comfortable at rest. Ordinary physical activity causes undue dyspnea or fatigue, chest pain or near-syncope.
  Class III: Patients with marked limitation of physical activity. They are comfortable at rest. Less than ordinary physical activity causes undue dyspnea or fatigue, chest pain or near-syncope.
  Participants
    Class I | 0
    Class II | 4
    Class III | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline of Plasma Estradiol Levels
Description: Plasma estradiol levels are obtained and measured from blood samples collected from each participant.
  Difference in change from baseline to 9 weeks in plasma estradiol levels
Time Frame: Baseline to 9 weeks
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Fulvestrant
Number analyzed (Participants) | 5
pg/ml | -1.26 [-1.7 to -0.26]

2. Primary Outcome: Change From Baseline of Tricuspid Annular Plane Systolic Excursion (TAPSE)
Description: Measure obtained from echocardiogram completed on participants Difference in change from baseline to 9 weeks in TAPSE
Time Frame: Baseline to 9 weeks
Measure: Median (Inter-Quartile Range); unit: millimeter
Arm/Group | Fulvestrant
Number analyzed (Participants) | 5
millimeter | 2 [-3 to 5.5]

3. Primary Outcome: Change From Baseline of Six Minute Walk Distance
Description: Measure obtained from six minute walk test completed by participants Difference in change from baseline to 9 weeks in the six minute walk test distance
Time Frame: Baseline to 9 weeks
Measure: Median (Inter-Quartile Range); unit: meters
Arm/Group | Fulvestrant
Number analyzed (Participants) | 5
meters | 31 [10 to 32]

4. Primary Outcome: Change From Baseline of Plasma NT-proBNP Level
Description: Plasma NT-proBNP levels are obtained and measured from blood samples collected from each participant.
  Difference in change from baseline to 9 weeks in plasma NT-proBNP levels
Time Frame: Baseline to 9 weeks
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Fulvestrant
Number analyzed (Participants) | 5
pg/ml | 42.1 [6.7 to 114]

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Fulvestrant
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 5/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fulvestrant (N=5)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Injection Site Pain (General disorders) | 1 (1)
Hot flashes (Nervous system disorders) | 1 (1)
Shoulder pain (General disorders) | 1 (1)
Worsened dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Joint pain (General disorders) | 1 (1)
Worsening hemodynamics (Cardiac disorders) | 1 (1)
Increased NT-proBNP level (Cardiac disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Small size Open-label and uncontrolled design, making it difficult to directly attribute the findings to the study intervention Short duration of the study may have affected the results

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-18): https://cdn.clinicaltrials.gov/large-docs/44/NCT02911844/Prot_SAP_000.pdf